CLINICAL TRIAL: NCT01713803
Title: Evaluation of BEMA® Buprenorphine NX for Buprenorphine Induction of Opioid Dependent Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA did not require a clinical trial for indication.
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Other Study IDs: BNX-350
Record Dates: First submitted 2012-10-19; First posted 2012-10-25 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Buprenorphine and naloxone
- buprenorphine and nalaxone (Experimental)
  Interventions: Drug: Buprenorphine and naloxone

INTERVENTIONS:
Drug: Buprenorphine and naloxone

SUMMARY:
This is a randomized, double blind, placebo controlled study in opioid dependent subjects. Subjects meeting entry criteria will be treated with multiple doses of B-BNX or B-Placebo, with non-responders rescued within 6 hours. Open treatment B-BNX will be administered as follow-up therapy. Clinical efficacy assessments include the clinical opioid withdrawal scale (COWS), subject-rated assessments, and a urine drug screen.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to any study procedure being performed
* Subject is a male or non-lactating female with a negative urine pregnancy test
* Subject is aged 18 to 65 years, inclusive
* Current diagnosis of opioid dependence or addiction per the Diagnostic and Statistical Manual of Mental Disorders - 4th edition (text revision) (DSM-IV-TR) criteria including physical dependence on opioids
* Daily short-acting opiate use of at least 60 mg morphine equivalent no opioid use for at least 12 hours prior to Screening with positive opiate result on urine drug screen
* Clinical opioid withdrawal scale (COWS) score ≥9
* Subject is in good general health in the judgment of the Investigator as determined from the physical and oral examination findings.

Exclusion Criteria:

* Use of a long-acting opioid within the last 72 hours
* Use of an investigational drug or device within the last 30 days
* History of hypersensitivity, allergy, or intolerance to buprenorphine, naloxone, or related drugs
* Immediate suicidal risk, as determined by meeting any of the following:

  1. History of suicidal ideation ≤ 3 months prior to Baseline with a score of 4 (intent to act) or 5 (specific plan and intent) on the eC-SSRS
  2. History of suicidal behavior ≤1 year prior to Baseline (actual attempt, interrupted attempt, aborted attempt and/or preparatory acts/behavior) on the eC-SSRS
* A history or current evidence of any clinically significant disorder or any other condition which in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
The mean change in clinical opioid withdrawal scale (COWS) total score from Baseline to 6 hours following the initial dose

SECONDARY OUTCOMES:
The percentage of subjects with a negative result on the urine drug screen at Day 7
The percentage of subjects with a clinical opioid withdrawal scale (COWS) total score ≤4 at 6 hours after the initial study drug dose

CONTACTS AND LOCATIONS:
Locations (1):
- Birmingham, Alabama, United States